CLINICAL TRIAL: NCT02691793
Title: Study to Evaluate the Safety and Efficacy of Sunitinib, in Subject With Refractory Solid Tumors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Seung tae Kim,PhMD, Principal Investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-02-098
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Refractory Solid Tumors
MeSH Terms: interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- sunitinib (Experimental): sunitinib 50 mg will be administered orally daily
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — sunitinib 37.5mg QD

SUMMARY:
This study is a single arm, pilot study of Sunitinib in patient with RET fusion positive, FGFR2 fusion/FGFR mutation Refractory solid tumor and/or specific sensitivity to Sunitinib by Avatar scan that has progressed following standard therapy or that has not responded to standard therapy or for which there is no standard therapy.

To investigate the efficacy and safety of Sunitinib in patient with Refractory solid tumor.

ELIGIBILITY:
Inclusion Criteria:

* Provision of fully informed consent prior to study specific procedures.
* Patients must be >= 19 years of age
* RET fusion positive or FGFR2 fusion/other FGFR mutation Refractory solid tumor and/or specific sensitivity to Sunitinib by Avatar scan that has progressed following standard therapy or that has not responded to standard therapy or for which there is no standard therapy.
* ECOG Performance status0-2
* Have measurable or evaluated disease based on RECIST 1.1 as determined by investigator.
* Adequate Organ Function Laboratory values

  * Absolute neutrophil count >= 1.5 x 109/L, Hemoglobin >= 9g/dL, Platelets>=100 x 109/L Bilirubin <= 1.5 x upper limit of normal AST/ALT <= 2.5 X upper limit of normal(5.0 x upper limit of normal, for subject with liver metastases) Creatinine<= 1.5 X UNL
* Patients of child-bearing potential should be using adequate contraceptive measures should not be breast feeding and must have a negative pregnancy test prior to start of dosing
* Adequate heart function

Exclusion Criteria:

* Patients with second primary cancer, except:adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumor curatively treated with no evidence of disease for <= 5 years.
* Has known active central nervous system(CNS) metastases
* Has an active infection requiring systemic therapy
* Pregnancy or breast feeding
* Patients with cardiac problem
* Any previous treatment with sunitinib

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 24 months

SECONDARY OUTCOMES:
overall response rate | 24 months
Time to progression | 24 months
overall survival | 24 months
Number of subjects with adverse events as a measure of safety | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Seoul, Korea, Republic of, South Korea